CLINICAL TRIAL: NCT02712567
Title: A Continuation Study of TH-CR-406/SARC021 for the Remaining Subjects Enrolled in TH-CR-406/SARC021 in the US
Brief Title: SARC021C: A Continuation Study of TH-CR-406/SARC021
Status: No longer available | Type: Expanded Access
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Collaborators: Threshold Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: SARC021C
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — TH 302

INTERVENTIONS:
Drug: Th-302 — 300 mg/m2 IV on Days 1 and 8 of a 21-day cycle.

SUMMARY:
SARC021C is a nonrandomized, open-label, multicenter, continuation study designed to provide access to TH-302 for patients currently receiving and benefiting from single agent TH-302 therapy as part of the Phase III TH-CR-406/SARC021 study.

DETAILED DESCRIPTION:
The goal of this study is to provide continuation therapy with TH-302 to patients with soft tissue sarcomas who obtained response or stabilization of disease with prior treatment on TH-CR-406/SARC021 protocol. After written informed consent has been obtained and eligibility has been established, patients will receive the study drug as part of the continuation study. Patients will receive treatment on study as long as they have clinical benefit and do not experience unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee.
* Previously enrolled on the TH-CR-406/SARC021 protocol and benefiting from treatment.
* Study investigator deems continued participation is appropriate based on overall health of the patient.

Exclusion Criteria:

* Any of the criteria for study discontinuation are met.
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
* Unwillingness or inability to comply with the study protocol for any reason.

Sex: All
Age Groups: Child, Adult, Older Adult